CLINICAL TRIAL: NCT07100418
Title: A Multicenter, Randomized, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of HRS-7249 in Patients With Hyperlipidemia
Brief Title: A Clinical Study Evaluating the Efficacy and Safety of HRS-7249 in Treating Patients With Hyperlipidemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-7249-201
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-7249 Group (Experimental)
  Interventions: Drug: HRS-7249 Injection
- Sodium Chloride Injection Group (Placebo Comparator)
  Interventions: Drug: Sodium Chloride Injection

INTERVENTIONS:
Drug: HRS-7249 Injection — HRS-7249 injection.
  Arms: HRS-7249 Group
Drug: Sodium Chloride Injection — Sodium chloride injection.
  Arms: Sodium Chloride Injection Group

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of HRS-7249 for patients with hyperlipidemia, and to explore the reasonable dosage of HRS-7249 for patients with hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent.
2. Age ≥ 18 years old and < 80 years old.
3. Male or female.

Exclusion Criteria:

1. Acute pancreatitis within 3 months or within 4 weeks or planned for plasma exchange treatment.
2. Malignant tumors within 5 years.
3. Severe cardiovascular or cerebrovascular diseases.
4. Severe trauma or surgery within 6 months or severe infection within 3 months.
5. Previous diagnosed diseases affecting lipid levels.
6. Patients with unstable or severe diseases assessed as at risk by the investigator.
7. Uncontrolled hypertension.
8. Weight loss within 2 months or planned surgery causing unstable weight.
9. Uncontrolled diabetes.
10. Combined hyperthyroidism or hypothyroidism.
11. History of drug or alcohol abuse.
12. Significantly abnormal liver or kidney function.
13. Significantly abnormal blood routine.
14. Significantly abnormal thyroid function.
15. Participated in clinical research within 3 months.
16. Pregnant or lactating women, or refusing contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
The level of triglyceride (TG) | About 28 weeks.

SECONDARY OUTCOMES:
Adverse events (AEs) | About 48 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided